CLINICAL TRIAL: NCT04412395
Title: Clinical Assessment of Oral Lactoferrin as a Safe Antiviral and Immunoregulatory Therapy in Patients Diagnosed With COVID-19 Disease
Brief Title: Clinical Assessment of Oral Lactoferrin as a Safe Antiviral and Immunoregulatory in Treating COVID-19 Disease
Acronym: COVID-19_LF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Research Centre, Egypt (Other)
Collaborators: Egyptian Military Medical Services (Other Government)
Responsible Party: Principal Investigator, Rehab Ragab Hegazy, Assistant Professor, National Research Centre, Egypt
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COVID-19_LF
Record Dates: First submitted 2020-05-15; First posted 2020-06-02 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Corona Virus Infection; Middle East Respiratory Syndrome (MERS); Acute Respiratory Distress Syndrome; Coronavirus Infection; COVID-19; SARS-CoV 2
Keywords: Lactoferrin; Apolactoferrin; Immuno-modulatory; Cytokine-storm; Antiviral; 2019nCoV; 2019 new coronavirus (2019nCoV); Middle East Respiratory Syndrome (MERS); Acute Respiratory Distress Syndrome (ARDS); COVID-19; SARS-CoV 2
MeSH Terms: conditions — Coronavirus Infections; Respiratory Distress Syndrome; COVID-19; Cytokine Release Syndrome | interventions — Lactoferrin; apolactoferrin

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 01 (SOC + Lactoferrin 1200 mg QID) (Active Comparator): Patients randomized to this group will receive two 600 mg Lactoferrin tablets QID plus the Standard of Care (SOC) treatment(s).
  Interventions: Dietary Supplement: Lactoferrin (Apolactoferrin)
- Arm 02 (SOC + Placebo QID) (Placebo Comparator): Patients randomized to this group will receive two placebo tablets QID plus the SOC treatment(s).
  Interventions: Drug: Placebo of excipient(s) will be administered

INTERVENTIONS:
Dietary Supplement: Lactoferrin (Apolactoferrin) — Apolactoferrin is an iron-free Lactoferrin (with very low iron saturation). Lactoferrin (Lf) is a natural glycoprotein that is found predominantly in milk. Lf represents a known component of the innate immune system present in neutrophil-specific granules and broadly distributed within the body fluids and exocrine secretions.
  Arms: Arm 01 (SOC + Lactoferrin 1200 mg QID)
Drug: Placebo of excipient(s) will be administered — Placebo of the equivalent excipient will be administered to placebo group
  Other Names: excipient(s)
  Arms: Arm 02 (SOC + Placebo QID)

SUMMARY:
The aim of the study is to clinically use bovine Lf as a safe antiviral adjuvant for treatment and to assess the potential in reducing mortality and morbidity rates in COVID-19 patients. The study was approved by the ethical committee of the Egyptian Center for Research and Regenerative Medicine in 11-5-2020.

DETAILED DESCRIPTION:
The World Health Organization (WHO) declared the coronavirus (SARS-CoV-2, COVID-19) outbreak a Public Health Emergency of International Concern with a pandemic spread. The situation is rapidly evolving, which raises the approach of reproposing already approved drugs to meet the emerging challenge and to save time and money. Lactoferrin (Lf) is a natural glycoprotein that broadly distributed within the body fluids and found predominantly in milk. It represents a known component of the innate immune system. The antiviral activity of Lf has been reported against many viruses, including SARS-CoV-1, through blocking the viral receptors on the host cells preventing them from entry and replication. Markedly, data reveals that Lf interacts with Heparan Sulfate Proteoglycans (HSPGs) and Angiotensin Converting Enzyme 2 (ACE2) receptors that are reported as SARS-CoV-2-binding sites to enter the host cell, suggesting a potential significance of Lf as an antiviral against SARS-CoV-2. Moreover, the immunoregulatory effects of Lf can protect against the cytokine-storm and thrombotic complications that result from the COVID-19-induced over-stimulated inflammatory response and exaggerated immune reactions. In addition, Lf can decrease the free iron toxicity caused by the virus as it has a strong iron chelating ability. Lf is a safe approved food supplement that is available in the markets for enhancement of immunity and for treatment of anemia. The aim of this study is to perform a randomized, double-blind, placebo-controlled, two arms, clinical trial to assess oral enteric-coated tablet of bovine apolactoferrin (the low iron-content form of Lf) as a safe antiviral and immunoregulatory therapy in patients diagnosed with COVID-19 disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients tested positive (PCR) for SARS-CoV-2 and clinically symptomatic.
* Adult patients with age >18 years.
* Patients willing and able to sign the study informed consent form.

Exclusion Criteria:

* Critically severe disease patients (having Respiratory failure requiring mechanical ventilation, or signs of septic shock or multiple organ failure requiring ICU admission).
* Patients who are unconscious
* Patients who have convulsions
* Patients suffering from central cyanosis with SPO2< 90% (for asthmatic patients with SPO2<88%)
* Pregnant or lactating women
* Patients with a known history of pro-inflammatory diseases (patients with autoimmune diseases, patients receiving chemotherapy for cancer, patients with malabsorption, patients with inflammatory bowel disease, Crohn's disease or ulcerative colitis).
* History or suspected immunosuppressive or immunodeficient state including HIV infection, or chronic immunosuppressant medication (more than 14 days) within the past 3 months (inhaled and topical steroids are allowed).
* Patients with severe renal impairment (GFR <60 ml/min/1.73m2 as measured by the Cockcroft-Gault formula).
* Patient with severe hepatic impairment, biliary cirrhosis or cholestasis
* Patients who received immunoregulatory therapy within one month before the start of the study.
* Patients with Known or suspected allergy or any contraindications to Lactoferrin.
* Any condition, according to the judgment of the investigator, would interfere with the patient's ability to comply with all study requirements or that would place the patient at unacceptable risk by his/her participation in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Survival rate. | up to 8 weeks.
  Comparing the influence of the intervention on the Survival rate.
Rate of disease remission. | up to 4 weeks.
  For mild/moderate symptoms patients: fever, cough and other symptoms relieved with improved lung CT
  - For severe symptoms patients: fever, cough and other symptoms relieved with improved lung CT, and oxygen saturation by pulse oximetry (SPO2 )> 93% for nonasthmatic patients, and from 88-92% in asthmatic patients.
The number of patients with PCR negative results. | up to 4 weeks.
  Comparing the influence of the intervention on the PCR negative results.

SECONDARY OUTCOMES:
Mean change in the disease severity (clinical assessment). | up to 4 weeks.
  Recording the changes from severe to moderate or mild and the time taken.
Mean change in blood pressure. | up to 4 weeks.
  Recording the changes in blood pressure mmHg.
Mean change in heart beats. | up to 4 weeks.
  Recording the changes in heart rate in beat/second.
Mean change in body temperature. | up to 4 weeks.
  Recording the changes in body temperature in Celsius.
Mean change in body respiratory rate. | up to 4 weeks.
  Recording the changes in the respiratory rate in breath/minute.
Mean change in oxygen saturation. | up to 4 weeks.
  Recording the changes in arterial oxygen saturation in mmHg.
Mean change in the ratio in arterial oxygen partial pressure to fractional inspired oxygen (PF ratio). | up to 4 weeks.
  Recording the changes in the ratio of arterial oxygen partial pressure to fractional inspired oxygen (PF ratio).
Mean change in complete blood picture (CBC). | up to 4 weeks.
  Recording the changes in complete blood picture (CBC) in cells per liter.
Mean change in C reactive protein (CRP). | up to 4 weeks.
  Recording the changes in C reactive protein (CRP) in mg/L.
Mean change in erythrocyte sedimentation rate (ESR). | up to 4 weeks.
  Recording the changes in erythrocyte sedimentation rate (ESR) in mm/hr.
Mean change in D-dimer. | up to 4 weeks.
  Recording the changes in D-dimer in ng/mL.
Mean change in ferritin. | up to 4 weeks.
  Recording the changes in ferritin in ng/mL.
Mean change in liver Albumin. | up to 4 weeks.
  Recording the changes in liver Albumin in g/L.
Mean change in total and direct Bilirubin. | up to 4 weeks.
  Recording the changes in total and direct Bilirubin in mg/dL.
Mean change in prothrombin time (PT) and partial thromboplastin time (PTT ). | up to 4 weeks.
  Recording the changes in prothrombin time (PT), partial thromboplastin time (PTT ) in seconds and calculating International Normalized Ratio (INR).
Mean change in aspartate aminotransferase (AST). | up to 4 weeks.
  Recording the changes in aspartate aminotransferase (AST) in IU/L.
Mean change in Alanine Aminotransferase (ALT). | up to 4 weeks.
  Recording the changes in Alanine Aminotransferase (ALT) in IU/L.
Mean change in Blood Urea Nitrogen (BUN). | up to 4 weeks.
  Recording the changes in Blood Urea Nitrogen (BUN) in mg/dL.
Mean change in Serum Creatinine. | up to 4 weeks.
  Recording the changes in Serum Creatinine in mg/dL.
Mean change in Serum Creatinine clearance. | up to 4 weeks.
  Recording the changes in Serum Creatinine in ml/min.
Mean change in Glomerular filtration rate (GFR ). | up to 4 weeks.
  Recording the changes in Glomerular filtration rate (GFR ) ml/min/m2.
The mean change in serum interleukin-1 (IL-1). | up to 4 weeks.
  Recording the changes in interleukin-1 (IL-1) in pg/ml.
The mean change in serum interleukin-6 (IL-6). | up to 4 weeks.
  Recording the changes in interleukin-6 (IL-6) in pg/ml.
The mean change in serum interleukin-10 (IL-10). | up to 4 weeks.
  Recording the changes in interleukin-10 (IL-10) in pg/ml.
The mean change in serum tumor necrosis factor-alpha (TNF alpha). | up to 4 weeks.
  Recording the changes in tumor necrosis factor-alpha (TNF alpha) in ng/ml.
Mean changes in immunoglobulin G (IgG). | up to 4 weeks.
  Recording the changes in immunoglobulin G (IgG) in ng/ml.
Mean changes in immunoglobulin M (IgM). | up to 4 weeks.
  Recording the changes in immunoglobulin M (IgM) in ng/ml.
The mean change in PCR viral load. | up to 4 weeks.
  Recording the changes in PCR viral load in copies/mL.
Mean change in lung CT manifestation. | up to 4 weeks.
  Recording the changes in lung CT.
Nature and severity of Adverse Events. | up to 4 weeks.
  Recording any unexpected Adverse Events of the intervention.
Time for lung recovery. | up to 8 weeks.
  Recording the changes (the average time of lung imaging recovery), as assessed by lung CT.
The number of missed drug doses among each treatment group. | up to 4 weeks.
  Recording the changes the event of missed drug doses.

CONTACTS AND LOCATIONS:
Overall Officials: Rehab Hegazy, PhD, Study Director — National Research Center
Locations (4):
- Egypt (4):
  - National Research Center, Egypt (Clinical and Molecular Pharmacology), Cairo, Giza Governorate
  - Clinmax CRO (Clinical Research Organization), Cairo
  - Clinical Trial Unit National Research Center, Cairo
  - Egyptian Military Medical Services (Hospitals), Cairo

IPD SHARING:
Plan to Share IPD: Yes
Not yet decided.
Time Frame: within 6 month
Access Criteria: all valid data